CLINICAL TRIAL: NCT03593239
Title: A Ten Sequence, Open Label, Randomized Crossover Study Comparing Nicotine Pharmacokinetics of JUUL 1.7% and JUUL 5% Nicotine Salt Based Electronic Nicotine Delivery System (ENDS Products), in Healthy Adult Smokers
Brief Title: Comparing the Pharmacokinetics of Nicotine Salt Based ENDS in Healthy Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juul Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PROT-00008 / v2.1
Record Dates: First submitted 2018-06-01; First posted 2018-07-20 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Nicotine Dependence; Nicotine Dependence, Cigarettes; Tobacco Use; Tobacco Smoking
Keywords: Electronic Nicotine Delivery System; Combustible Cigarettes; Nicotine
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use; Tobacco Smoking; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- Tobacco flavored JUUL 1.7% ENDS (Experimental): Tobacco flavored JUUL 1.7% ENDS (10 puffs)
  Interventions: Other: Tobacco flavored JUUL 1.7% ENDS
- Tobacco flavored JUUL 5% ENDS (Experimental): Tobacco flavored JUUL 5% ENDS (10 puffs)
  Interventions: Other: Tobacco flavored JUUL 5% ENDS
- Mint flavored JUUL 1.7% ENDS (Experimental): Mint flavored JUUL 1.7% ENDS (10 puffs);
  Interventions: Other: Mint flavored JUUL 1.7% ENDS
- Mint flavored JUUL 5% ENDS (Experimental): Mint flavored JUUL 5% ENDS (10 puffs)
  Interventions: Other: Mint flavored JUUL 5% ENDS
- Fruit Medley flavored JUUL 1.7% ENDS (Experimental): Fruit Medley flavored JUUL 1.7% ENDS (10 puffs)
  Interventions: Other: Fruit Medley flavored JUUL 1.7% ENDS
- Fruit Medley flavored JUUL 5% ENDS (Experimental): Fruit Medley flavored JUUL 5% ENDS (10 puffs)
  Interventions: Other: Fruit Medley flavored JUUL 5% ENDS
- Crème brulee flavored JUUL 1.7% ENDS (Experimental): Crème brulee flavored JUUL 1.7% ENDS (10 puffs)
  Interventions: Other: Crème brulee flavored JUUL 1.7% ENDS
- Crème brulee flavored JUUL 5% ENDS (Experimental): Crème brulee flavored JUUL 5% ENDS (10 puffs)
  Interventions: Other: Crème brulee flavored JUUL 5% ENDS
- JUUL 1.7% ENDS 10 puffs vs. ad lib puffs (Experimental): Tobacco flavoured JUUL 1.7% ENDS products 10 puffs versus ad libitum puffs
  Interventions: Other: JUUL 1.7% ENDS 10 puffs vs. ad lib puffs
- JUUL 5% ENDS 10 puffs vs. ad lib puffs (Experimental): Tobacco flavoured JUUL 5% ENDS products 10 puffs versus ad libitum puffs
  Interventions: Other: JUUL 5% ENDS 10 puffs vs. ad lib puffs

INTERVENTIONS:
Other: Tobacco flavored JUUL 1.7% ENDS — Treatment with Tobacco flavored JUUL 1.7% ENDS (10 puffs)
  Arms: Tobacco flavored JUUL 1.7% ENDS
Other: Tobacco flavored JUUL 5% ENDS — Treatment with Tobacco flavored JUUL 5% ENDS(10 puffs)
  Arms: Tobacco flavored JUUL 5% ENDS
Other: Mint flavored JUUL 1.7% ENDS — Treatment with Mint flavored JUUL 1.7% ENDS(10 puffs)
  Arms: Mint flavored JUUL 1.7% ENDS
Other: Mint flavored JUUL 5% ENDS — Treatment with Mint flavored JUUL 5% ENDS(10 puffs)
  Arms: Mint flavored JUUL 5% ENDS
Other: Fruit Medley flavored JUUL 1.7% ENDS — Treatment with Fruit Medley flavored JUUL 1.7% ENDS(10 puffs)
  Arms: Fruit Medley flavored JUUL 1.7% ENDS
Other: Fruit Medley flavored JUUL 5% ENDS — Treatment with Fruit Medley flavored JUUL 5% ENDS(10 puffs)
  Arms: Fruit Medley flavored JUUL 5% ENDS
Other: Crème brulee flavored JUUL 1.7% ENDS — Treatment with Crème brulee flavored JUUL 1.7% ENDS(10 puffs)
  Arms: Crème brulee flavored JUUL 1.7% ENDS
Other: Crème brulee flavored JUUL 5% ENDS — Treatment with Crème brulee flavored JUUL 5% ENDS(10 puffs)
  Arms: Crème brulee flavored JUUL 5% ENDS
Other: JUUL 1.7% ENDS 10 puffs vs. ad lib puffs — Treatment with JUUL 1.7% ENDS 10 puffs vs. ad libitum puffs
  Arms: JUUL 1.7% ENDS 10 puffs vs. ad lib puffs
Other: JUUL 5% ENDS 10 puffs vs. ad lib puffs — Treatment with JUUL 5% ENDS 10 puffs vs. ad libitum puffs
  Arms: JUUL 5% ENDS 10 puffs vs. ad lib puffs

SUMMARY:
A Ten Sequence, Open Label, Randomized Crossover Study Comparing Nicotine Pharmacokinetics of JUUL 1.7% and JUUL 5% Nicotine Salt Based ENDS Products, in Healthy Adult Smokers.

DETAILED DESCRIPTION:
E-cigarettes may be an acceptable alternative to traditional cigarette smoking. In utilizing vaporization rather than combustion, the generation and inhalation of smoke and carbon monoxide (CO) may be reduced or avoided. JUUL has developed several nicotine based liquid blends for use in e-cigarettes. This study will provide an understanding of the levels of nicotine obtained with use of the company's 1.7% and 5% ENDS products.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 60 years of age inclusive.
* Current smoker or e-cigarette user:
* Able to participate, and willing to give written informed consent and to comply with the ° study restrictions.

Exclusion criteria:

* Clinically significant abnormality on screening ECG.
* Sustained blood pressure recordings at screening of < 90 mmHg or > 150 mmHg for systolic blood pressure, or < 50 mmHg or > 90 mmHg for diastolic blood pressure.
* Sustained resting heart rate of > 100 or < 40 beats per minute at screening.
* Positive result for urine drugs of abuse test or alcohol breath test at screening.
* Clinically significant abnormality in laboratory test results at screening, in the opinion of the Investigator.
* Positive urine pregnancy test at screening or Assessment Days in female subjects of child bearing potential.
* Any clinically significant concomitant disease or conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Compare nicotine pharmacokinetics(PK) in smokers and e-cigarette users measuring Time to Maximum Concentration(Tmax) | 38 Days
  Compare nicotine pharmacokinetics (PK) in smokers and e-cigarette users, obtained with:
  Tobacco flavored JUUL 1.7% ENDS (10 puffs); Tobacco flavored JUUL 5% ENDS (10 puffs); Mint flavored JUUL 1.7% ENDS (10 puffs); Mint flavored JUUL 5% ENDS (10 puffs); Fruit Medley flavored JUUL 1.7% ENDS (10 puffs); Fruit Medley flavored JUUL 5% ENDS (10 puffs); Crème brulee flavored JUUL 1.7% ENDS (10 puffs); Crème brulee flavored JUUL 5% ENDS (10 puffs).
Compare nicotine pharmacokinetics(PK) in smokers and e-cigarette users measuring Concentration Maximum (Cmax) | 38 Days
  Compare nicotine pharmacokinetics (PK) in smokers and e-cigarette users, obtained with:
  Tobacco flavored JUUL 1.7% ENDS (10 puffs); Tobacco flavored JUUL 5% ENDS (10 puffs); Mint flavored JUUL 1.7% ENDS (10 puffs); Mint flavored JUUL 5% ENDS (10 puffs); Fruit Medley flavored JUUL 1.7% ENDS (10 puffs); Fruit Medley flavored JUUL 5% ENDS (10 puffs); Crème brulee flavored JUUL 1.7% ENDS (10 puffs); Crème brulee flavored JUUL 5% ENDS (10 puffs).
Compare nicotine pharmacokinetics(PK) in smokers and e-cigarette users measuring Cmax-baseline and Area Under the Curve ( AUC) 1hour | 38 Days
  Compare nicotine pharmacokinetics (PK) in smokers and e-cigarette users, obtained with:
  Tobacco flavored JUUL 1.7% ENDS (10 puffs); Tobacco flavored JUUL 5% ENDS (10 puffs); Mint flavored JUUL 1.7% ENDS (10 puffs); Mint flavored JUUL 5% ENDS (10 puffs); Fruit Medley flavored JUUL 1.7% ENDS (10 puffs); Fruit Medley flavored JUUL 5% ENDS (10 puffs); Crème brulee flavored JUUL 1.7% ENDS (10 puffs); Crème brulee flavored JUUL 5% ENDS (10 puffs).
Compare nicotine pharmacokinetics(PK) in smokers and e-cigarette users measuring AUC1hour-baseline of nicotine | 38 Days
  Compare nicotine pharmacokinetics (PK) in smokers and e-cigarette users, obtained with:
  Tobacco flavored JUUL 1.7% ENDS (10 puffs); Tobacco flavored JUUL 5% ENDS (10 puffs); Mint flavored JUUL 1.7% ENDS (10 puffs); Mint flavored JUUL 5% ENDS (10 puffs); Fruit Medley flavored JUUL 1.7% ENDS (10 puffs); Fruit Medley flavored JUUL 5% ENDS (10 puffs); Crème brulee flavored JUUL 1.7% ENDS (10 puffs); Crème brulee flavored JUUL 5% ENDS (10 puffs).

SECONDARY OUTCOMES:
Change in Pre and Post exhaled carbon monoxide (CO) values for each subject and Test Product. | 38 Days
  Change in Pre and Post exhaled carbon monoxide (CO) values for each subject and Test Product.
To compare user satisfaction measures of each Test Product when consumed by smokers and e-cigarette users. | 38 Days
  Measure of subjective product evaluation using the "modified Product Evaluation Scale (mPES)" Change in Evaluation; Scale: 1 = not at all, 2 = very little, 3 = a little, 4 = moderately, 5 = a lot, 6 = quite a lot, 7 = extremely
  Four multi-item subscales will be derived from "Satisfaction" (items 1, 2, 3, and 12); "Psychological Reward" (items 4 through 8); "Aversion" (items 9, 10, 16, and 18); and "Relief" (item 11, 13, 14, 15, and reversed for item 19) and single items 17 and 20 will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Wynne, MD, Principal Investigator — Christchurch Clinical Studies Trust Ltd
Locations (1):
- Christchurch Clinical Studies Trust Ltd, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No